CLINICAL TRIAL: NCT02336477
Title: Efficacy and Safety of Mexiletine in Non-dystrophic Myotonias
Brief Title: Mexiletine and Non Dystrophic Myotonias
Acronym: MYOMEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P091101
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Non-dystrophic Myotonias; Paramyotonia Congenita; Myotonia Congenita
Keywords: non-dystrophic myotonias; paramyotonia congenita; myotonia congenita; Mexiletine; Randomized clinical trial
MeSH Terms: conditions — Myotonic Disorders; Myotonia Congenita | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mexiletine / Placebo
  Interventions: Drug: Mexiletine; Drug: placebo
- 2 (Experimental): Placebo / Mexiletine
  Interventions: Drug: Mexiletine; Drug: placebo

INTERVENTIONS:
Drug: Mexiletine — * Blisters of 10 capsules of 200 mg mexiletine hydrochloride.
  * Patients will receive gradual dose of the treatment as it would be done in clinical practice.
  * Mexiletine will be started at 200 mg / day (1 capsule to be taken at the beginning of the meal) and will be increased by 200mg every 3 days to reach a maximum of 600mg / day in 3 taken in 1 week.
  * The duration of each treatment period is 18 days minimum (maximum 22 days).
Drug: placebo

SUMMARY:
Treatment strategies in non-dystrophic myotonias are based on selective case reports, clinical experience and theoretical benefit. Presently, the most promising antimyotonic medication is mexiletine (MEX) but its manufacturing was stopped. The proposed randomized, double-blind, placebo-controlled, crossover trial is designed to:

1. study the safety and efficacy of mexiletine for the treatment of non-dystrophic myotonias
2. validate electromyographic tests as a standardized outcome measure of myotonia
3. assess the reliability and validity of a new clinical rating scale for myotonia

DETAILED DESCRIPTION:
A. Specific aims

Treatment strategies in non-dystrophic myotonias are based on selective case reports, clinical experience and theoretical benefit. Presently, the most promising antimyotonic medication is mexiletine (MEX) but its manufacturing was stopped. The proposed randomized, double-blind, placebo-controlled, crossover with wash-out trial is designed to:

* study the safety and efficacy of mexiletine for the treatment of non-dystrophic myotonias
* validate electromyographic tests as a standardized outcome measure of myotonia
* assess the reliability and validity of a new clinical rating scale for myotonia

B. Research design Because of their differing phenotypes, 12 Paramyotonia Congenita and 12 Myotonia Congenita subjects will be enrolled in a stratified trial

C. Outcome variables

1. primary outcome variable: the score of stiffness severity on a self-assessment scale (100 mm VAS) measured at baseline, at the end of phase I and phase II.
2. secondary outcome measures:

   * of efficacy:

     * standardized EMG measures after repetitive short exercise test at cold and long exercise test
     * chair test: time needed to stand up from a chair, walk around it and sit down again
     * severity and disability scale of myotonia to be validated)
     * quality of life scale (INQOL)
     * rate of drop-outs
   * of safety:

     * adverse event frequency and severity
     * EKG

D. Perspectives

It is anticipated that the trial will:

1. provide data that justify recommendations for treatment strategies for myotonic patients
2. provide data to justify AFSAPPS regulatory approval of mexiletine for treatment of myotonia in order to guarantee the availability of the drug for patients
3. develop standardized diagnostic and treatment assessment for non-dystrophic myotonias

ELIGIBILITY:
Inclusion criteria :

* Genetically definite MC and PC.
* Male and female participants, age between 18 and 65 who are able to comply with the study conditions.
* Participants who experience myotonic symptoms severe enough to justify treatment.

The severity will be evaluated on:

* Clinical criteria: myotonia is considered as severe if it involves at least two segments (upper limb, lower limb or face)
* Disabling criteria: myotonia is considered severe if patients notice impacts on at least 3 of the 7 daily activities listed in the disabling section of the clinical myotonia scale (Annex 2).

Thus, patients who experience myotonic symptoms severe enough to justify treatment are those with myotonia that involves at least two segments and that have an impact on at least 3 daily activities.

* Participants who are drug naive or those who receiving mexiletine at Effective dosage and agreeing to stop treatment at least four days before inclusion .
* Pregnancy: Women: non-childbearing potential (i.e., postmenopausal or Surgically sterile) or must use a medically accepted contraceptive regimen; a pregnancy test will ensure that they are not pregnant.
* Normal cardiac exam performed by a cardiologist including EKG, and Cardiac ultrasound (if not done within 3 months before trial).

Exclusion criteria :

* Intercurrent event which could interfere with the muscle function (infection,trauma, fracture, …)
* Coincidental renal, hepatic, respiratory, thyroid, other neuromuscular disease or heart disease that will contraindicate mexiletine or interfere with clinical evaluation.
* Use of any of the following medications that can interfere with muscle function :diuretics, anti epileptics (sodium channel blockers), antiarrhythmics, corticosteroids, beta-blockers,
* Allergy to mexiletine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
score of stiffness severity on a self-assessment scale (100 mm VAS) | 18 days

SECONDARY OUTCOMES:
standardized EMG measures after repetitive short exercise test at cold and long exercise test | 18 days
chair test: time needed to stand up from a chair, walk around it and sit down again | 18 days
severity and disability scale of myotonia to be validated | 18 days
quality of life scale (INQOL) | 18 days
CGI efficacy (Clinical Global Impression- Efficacy index) | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Fontaine, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; Savine Vicart, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetriere, Paris, France